CLINICAL TRIAL: NCT00795808
Title: Multi-Centre Randomised Controlled Trial of the Effectiveness of Metformin and Clomiphene Citrate for Treating Anovulatory Infertility in Women With Polycystic Ovary Syndrome
Brief Title: PCOSMIC Trial - PolyCystic Ovary Syndrome, Metformin for Infertility With Clomiphene
Acronym: PCOSMIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Auckland Medical Research Foundation (Other); Mercia Barnes Trust of the Royal Australian and New Zealand College of Obstetricians and Gynaecologists (Other)
Responsible Party: Associate Professor Neil Johnson, University of Auckland, Fertility Plus and Repromed Auckland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UAuckland
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; PCOS; Anovulation; Infertility; Anovulatory polycystic ovary syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation; Infertility | interventions — Metformin; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMI > 32 (Experimental): Women with BMI > 32
  Interventions: Drug: Metformin; Drug: Placebo
- BMI </= 32 (Experimental): Women with BMI </= 32
  Interventions: Drug: Metformin + Clomiphene; Drug: Metformin; Drug: Clomiphene

INTERVENTIONS:
Drug: Metformin — 500mg tds for 6 months
  Arms: BMI > 32
Drug: Placebo — One tablet tds for 6 months
  Arms: BMI > 32
Drug: Metformin + Clomiphene — 500mg tds + Ovulatory dose for 6 months
  Arms: BMI </= 32
Drug: Metformin — 500mg tds for 6 months
  Arms: BMI </= 32
Drug: Clomiphene — Ovulatory dose for 6 months
  Arms: BMI </= 32

SUMMARY:
1. Metformin increases the pregnancy rate when added to the standard treatment of anovulatory polycystic ovary syndrome (PCOS).
2. Metformin in combination with clomiphene, is more effective than clomiphene alone or metformin alone improves fertility outcomes in women with PCOS of reasonably healthy body weight (BMI </= 32).
3. Metformin improves fertility outcomes in women with BMI > 32 with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Women between the age of 18 and 39 years inclusive.
* Anovulatory infertility of duration at least 12 months.
* Polycystic ovary syndrome, based on Rotterdam consensus criteria.
* Normal serum prolactin, thyroid function and 17-hydroxyprogesterone.
* Normal serum prolactin, thyroid function and 17-hydroxyprogesterone;

Exclusion Criteria:

* Presence of any other significant infertility factor including male factor, known tubal disease or history of an ectopic pregnancy, known endometriosis affecting the fallopian tubes or ovaries.
* Already taking oral hypoglycaemics.
* Diabetics receiving treatment.
* Renal impairment
* Chronic hepatic disease
* Cardiac Disease
* Alcohol dependency
* Pre-disposition to lactic acidosis
* Previous ovarian drilling procedure, gonadotrophin injection therapy, IUI (intrauterine insemination) or IVF ( in vitro fertilisation).
* For those women who have had previous fertility treatment, the following would be excluded:

  * Women who have had > 5 cycles of clomiphene citrate
  * Women who have had > 5 months metformin treatment previously
  * Women who have proven to be resistant to 100mg or more of clomiphene citrate.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2003-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | within 6 calendar months of randomisation

SECONDARY OUTCOMES:
Live birth
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Neil P Johnson, FRANZCOG, Principal Investigator — University of Auckland, fertility Plus & Repromed Auckland
Locations (1):
- University of Auckland, Auckland, New Zealand

REFERENCES:
- [Derived] Johnson NP, Stewart AW, Falkiner J, Farquhar CM, Milsom S, Singh VP, Okonkwo QL, Buckingham KL; REACT-NZ (REproduction And Collaborative Trials in New Zealand), a multi-centre fertility trials group. PCOSMIC: a multi-centre randomized trial in women with PolyCystic Ovary Syndrome evaluating Metformin for Infertility with Clomiphene. Hum Reprod. 2010 Jul;25(7):1675-83. doi: 10.1093/humrep/deq100. Epub 2010 Apr 30. PMID 20435692